CLINICAL TRIAL: NCT01274013
Title: A Pilot Study on Vitamin D Deficiency in Subjects With Chronic Hepatitis C Compared to Healthy Volunteers
Brief Title: Vitamin D Deficiency in Subjects With Chronic Hepatitis C Compared to Healthy Volunteers
Status: Withdrawn | Type: Observational
Why Stopped: Non Hep C study arm has been completed, Hep C study arm has not been completed.
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: ARI-1280-HEPC
Record Dates: First submitted 2011-01-07; First posted 2011-01-11 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C; Chronic Hepatitis C; Vitamin D; Vitamin D deficiency
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Study Group: Individuals with chronic Hepatitis C
- Control Group: Healthy individuals

SUMMARY:
The objective of this study is to assess the prevalence of vitamin D deficiency in patients with chronic Hepatitis C compared to a matched control group of healthy individuals in the Sioux Falls area. It is the hypothesis of this study that vitamin D deficiency is more common in patients with chronic Hepatitis C compared to the healthy control group.

DETAILED DESCRIPTION:
In this study, we will measure vitamin D levels in patients with chronic Hepatitis C and healthy individuals. This study will be important to assess vitamin D inadequacy in patients with chronic Hepatitis C and healthy individuals in this area.

ELIGIBILITY:
Inclusion Criteria for Study Group:

* Men and women between the ages of 25 and 55
* Diagnosis of chronic hepatitis C

Exclusion Criteria for Study Group:

* Taking a vitamin D supplement (by itself or as part of a multivitamin), a calcium supplement and/or biphosphonates
* Has acute hepatitis C infection
* Has chronic hepatitis B infection
* Had gastric bypass surgery
* Has chronic kidney disease

Inclusion Criteria for Control Group:

* Men and women between the ages of 20 and 60
* Has a body mass index (BMI) between 20 and 35

Exclusion Criteria for Study Group:

* Taking a vitamin D supplement (by itself or as part of a multivitamin), a calcium supplement and/or biphosphonates
* Has any significant illness or medical problem that is not under control or being controlled by medication
* History of hepatitis or abnormal liver chemistry tests
* History of intravenous drug use

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This is a comparison study between two different populations: a study group and a control group. The study group will consist of fifty individuals with a diagnosis of chronic Hepatitis C. The control group will consist of fifty individuals who are considered to be generally healthy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
The Vitamin D levels of the 100 subjects will be statistically analyzed as the primary variable and correlated with the rest of the variables via ANOVA and meta-analysis | Initial clinic visit
  This research study consists of a single clinic visit. After study subjects have completed the informed consent process and are determined to meet study eligibility, a blood sample will be collected. Values from these lab samples will be compared between study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Hesham Elgouhari, MD, Principal Investigator — Avera McKennan Hospital & University Health Center
Locations (1):
- Avera Research Institute, Sioux Falls, South Dakota, United States

REFERENCES:
- [Background] Peterlik M, Cross HS. Vitamin D and calcium deficits predispose for multiple chronic diseases. Eur J Clin Invest. 2005 May;35(5):290-304. doi: 10.1111/j.1365-2362.2005.01487.x. PMID 15860041
- [Background] DeLuca HF. Overview of general physiologic features and functions of vitamin D. Am J Clin Nutr. 2004 Dec;80(6 Suppl):1689S-96S. doi: 10.1093/ajcn/80.6.1689S. PMID 15585789
- [Background] Nagpal S, Na S, Rathnachalam R. Noncalcemic actions of vitamin D receptor ligands. Endocr Rev. 2005 Aug;26(5):662-87. doi: 10.1210/er.2004-0002. Epub 2005 Mar 29. PMID 15798098
- [Background] Fisher L, Fisher A. Vitamin D and parathyroid hormone in outpatients with noncholestatic chronic liver disease. Clin Gastroenterol Hepatol. 2007 Apr;5(4):513-20. doi: 10.1016/j.cgh.2006.10.015. Epub 2007 Jan 10. PMID 17222588
- [Background] Yano M, Ikeda M, Abe K, Dansako H, Ohkoshi S, Aoyagi Y, Kato N. Comprehensive analysis of the effects of ordinary nutrients on hepatitis C virus RNA replication in cell culture. Antimicrob Agents Chemother. 2007 Jun;51(6):2016-27. doi: 10.1128/AAC.01426-06. Epub 2007 Apr 9. PMID 17420205
- [Background] Boucher BJ, John WG, Noonan K. Hypovitaminosis D is associated with insulin resistance and beta cell dysfunction. Am J Clin Nutr. 2004 Dec;80(6):1666; author reply 1666-7. doi: 10.1093/ajcn/80.6.1666. No abstract available. PMID 15585785
- [Background] Dawson-Hughes B, Heaney RP, Holick MF, Lips P, Meunier PJ, Vieth R. Estimates of optimal vitamin D status. Osteoporos Int. 2005 Jul;16(7):713-6. doi: 10.1007/s00198-005-1867-7. Epub 2005 Mar 18. PMID 15776217